CLINICAL TRIAL: NCT00002287
Title: A Placebo-Controlled Trial to Evaluate Retrovir in Preventing Infection With the Human Immunodeficiency Virus (HIV) in Health Care Workers After Accidental Exposure
Brief Title: A Study of Retrovir in the Prevention of HIV Infection in Health Care Workers Accidentally Exposed to the Virus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 014I; 20
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-08

CONDITIONS: HIV Infections
Keywords: Health Manpower; Accidents, Occupational; Zidovudine
MeSH Terms: conditions — HIV Infections | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To evaluate the safety and effectiveness of Retrovir (AZT) when used as prophylaxis for health care workers at risk for HIV infection from exposure to HIV-contaminated blood or blood components.

ELIGIBILITY:
Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* A prior history of a malignancy other than cutaneous basal cell or cervical carcinomas.
* Other significant, chronic underlying medical illness which, in the physician's judgment, would impair study completion.
* Evidence of compromised bone marrow function (lab results) with a blood transfusion within the last month.
* Liver dysfunction as indicated by lab results.

Patients are excluded if there is a prior diagnosis of HIV infection by one of the following criteria:

* HIV antibody positive by ELISA and Western blot assays or by other certified test method. (Patients who are ELISA positive but Western blot or other confirmatory tests are negative may continue in study).
* HIV antigen positive.
* Clinical symptoms which lead to a diagnosis by a licensed physician of AIDS or AIDS related complex or AIDS-related dementia. Also excluded are individuals who have experienced similar HIV exposure as described in this protocol in the past month and individuals who have previously been enrolled in this study. The purpose of these exclusions is to eliminate possible seroconversion in an individual that could be attributed to HIV exposure other than the single exposure experienced just prior to entry into the study.

Prior Medication:

Excluded within 4 weeks of study entry:

* Any potentially myelosuppressive drug.
* Nephrotoxic agent.
* Other experimental therapy.

Exposure of a health care worker to HIV-contaminated blood or blood component within 5 days prior to beginning therapy, defined as one of the following:

* Penetrating wound from needle recently removed from patient or sample container (e.g., blood bag, blood tube) or from sharp object visibly contaminated with HIV-positive blood or blood component. In the case of needlesticks or cuts with sharp objects, blood or blood component must not have been exposed to the air for more than 1 hour. If actual infusion of blood occurs, the 1-hour time limit does not apply.
* Hypodermic needles should come in contact with the blood and blood component from an HIV source but need not be visibly contaminated with blood to be considered a source of contamination.
* Significant exposure to HIV-positive blood or blood component as the result of splash on abraded skin.
* Significant exposure to HIV-positive blood or blood component as the result of splash on mucous membranes.
* Participant must be able to give informed consent.

Active drug or alcohol abuse sufficient in the physician's opinion to prevent compliance with the study regimen.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Glaxo Wellcome Inc, Research Triangle Park, North Carolina, United States